CLINICAL TRIAL: NCT01513434
Title: Femoral Tunnel Position on Conventional MRI After Anterior Cruciate Ligament Reconstruction-Transtibial Technique Versus Transportal Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Police Hospital (Other Government)
Responsible Party: Principal Investigator, Jung Ho Noh, Principal investigator, National Police Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPH2008-004
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transtibial technique (Active Comparator): In anterior cruciate ligament reconstruction, femoral tunnel was made via tibial tunnel.
  Interventions: Procedure: transtibial technique; Procedure: anterior cruciate ligament reconstruction
- Transportal technique (Active Comparator): In anterior cruciate ligament reconstruction, femoral tunnel was made via anteromedial portal.
  Interventions: Procedure: Transportal technique; Procedure: anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: transtibial technique — Femoral tunnel was made via tibial tunnel in anterior cruciate ligament reconstruction.
  Arms: transtibial technique
Procedure: Transportal technique — Femoral tunnel was made via anteromedial portal in anterior cruciate ligament reconstruction.
  Other Names: anteromedial portal technique
  Arms: Transportal technique
Procedure: anterior cruciate ligament reconstruction — femoral and tibial tunneling graft fixation on the femoral side with endobutton and on the tibial side with post-tie and interference screw

SUMMARY:
The position of the femoral tunnel in anterior cruciate ligament (ACL) reconstruction has been assessed on three dimensional CT (3D-CT) scan or in cadaveric study. However, these methods have some issues; 3D-CT scan has a concern on radiation exposure and cadaveric study is not easily available nor an in vivo test. The purpose of this study is to compare the position of the femoral tunnel aperture on conventional MRI and the outcomes after single bundle ACL reconstruction using free tendon Achilles allograft between transportal technique and transtibial technique in active young men.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of anterior cruciate ligament rupture

Exclusion Criteria:

* female
* over 45 years old
* the subjects who had ACL reconstruction with graft other than Achilles allograft
* the subjects who had concomitant other ligament injuries on the same knee needing surgical treatment
* revision ACL reconstruction
* double bundle ACL reconstruction
* concomitant full thickness cartilage injury needing cartilage repairing surgery

Ages: 17 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Lysholm score | at least two years after surgery
  Lysholm score was superior in transportal technique to transtibial technique.
Position of femoral tunnel aperture | within one week after surgery
  The position of the femoral tunnel aperture with transportal technique was more posterior than that of transtibial technique.

CONTACTS AND LOCATIONS:
Locations (1):
- National Police Hospital, Seoul, South Korea